CLINICAL TRIAL: NCT06567223
Title: Effectiveness of Whole-Body Vibration Versus Rhythmic Auditory Stimulation on Spasticity, Balance, and Lower Limb Motor Function on Hemiplegic Stroke Patients
Brief Title: Effectiveness of WBV Versus RAS on Spasticity, Balance, and Lower Limb Motor Function on Hemiplegic Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/737
Record Dates: First submitted 2024-08-08; First posted 2024-08-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vibration Therapy (Experimental)
  Interventions: Procedure: Vibration Therapy
- Rhythmic auditory stimulation therapy. (Active Comparator)
  Interventions: Combination Product: Rhythmic auditory stimulation therapy.

INTERVENTIONS:
Procedure: Vibration Therapy — will receive the whole body vibration therapy. Patient will be ask to stand on the vibration plate in semi flexed knee position will 3 minute time of rest and therapy. It will be given for four weeks three days per week. Acceleration will be 18.0 meter per second square and frequency will be from 30 to 40 Hz. Intensity of the therapy will increase throughout all the sessions
  Arms: Vibration Therapy
Combination Product: Rhythmic auditory stimulation therapy. — will receive rhythmic auditory stimulation therapy. Rhythmic auditory stimulation will be given for 90 minutes along with 30 minutes of conventional physiotherapy. It will consist of 15 minutes of general body warming metronome rhythm which proceed towards RAS music based exercise of 60 minutes. This period also ends up with 15 minutes of relaxation exercise. Relaxing Music was provided through headphones having voice cancellation property for 15 min. The total session will be given three days per week for four weeks. Exercises such as lateral walking military march, anterior walking, one toe and one heel walking along with posterior walking through progression with the speed of the rhythm is done
  Arms: Rhythmic auditory stimulation therapy.

SUMMARY:
This study investigates the effectiveness of whole-body vibration (WBV) versus rhythmic auditory stimulation (RAS) on spasticity, balance, and lower limb motor function in hemiplegic stroke patients. The objective was to compare the two interventions to determine which provides greater benefits in stroke rehabilitation. Hemiplegic stroke patients were randomly assigned to either the WBV group, receiving whole-body vibration therapy, or the RAS group, undergoing rhythmic auditory stimulation sessions.

DETAILED DESCRIPTION:
The study measured spasticity using the Modified Ashworth Scale (MAS), balance with the Berg Balance Scale (BBS), and lower limb motor function through the Fugl-Meyer Assessment (FMA). Results indicated that both WBV and RAS significantly improved spasticity, balance, and lower limb motor function.

ELIGIBILITY:
Inclusion Criteria:

* Participant with Age from 40 to 60 years
* Both males and females
* Diagnosed CVA patients
* Chronic stage (after 6 months of onset
* Individuals with BBS score ≥ 20 ≤ 40
* FMI score up to 3(moderate assistance)
* Able to understand command
* Mini-Mental State Examination (MMSE) score of over 20

Exclusion Criteria:

* Systematic Disorder e.g. Rheumatoid arthritis
* Unstable Angina
* Coexisting physical impairments e.g. limb amputation
* Any previous history of neurological disease other than stroke e.g. Parkinson's
* Any previous history of fractures
* Hearing or perception deficits
* Individuals unable to adhere to the study protocol or attend scheduled follow-up visits.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 12 Months
  Modified Ashworth Scale is a scale which is used to assess spasticity in a patient. It is range from 0 to 4 where 0 shows no muscle tone with no range to 4 which shows maximum muscle tone with full range..
Berg balance scale | 12 months
  Balance was measured by using BBS which was created in 1989 to measure balance in the older people. The Berg balance scale 27 assesses practical balance performance on 14 things normal to everyday life. The scale comprises of 14 items, scored from 0 to 4, which are added to make an all-out score somewhere in the range of 0 and 56; a higher score shows better balance
Fugl-Meyer Assessment (FMA) | 12 months
  Fugl-Meyer Assessment (FMA) for Lower Limb. In order to assess the lower extremity motor control fugal Meyer assessment test which is a strokes specific test was used to assess the motor function balance and sensation in stroke patients. Its scoring is through 3 point ordinal scale where 2 is performed fully and 1 is performed partially. It has a maximum score of 34

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - Sehat Medical Complex, Hanjerwal, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No